CLINICAL TRIAL: NCT00829907
Title: Effect of ORM-12741 on Receptor Occupancy Studied by Positron Emission Tomography; an Open, Single Dose, Dose Ranging Study in Healthy Males
Brief Title: A PET Study With ORM-12741
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Orion Corporation, Orion Pharma (Aila Holopainen, Clinical Study Director), Clinical study management
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 3098005
Record Dates: First submitted 2008-12-11; First posted 2009-01-27 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Healthy volunteer study
MeSH Terms: interventions — ORM-12741

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Orm-12741
  Interventions: Drug: ORM-12741

INTERVENTIONS:
Drug: ORM-12741 — Single dose as a capsule, oral administration

SUMMARY:
The purpose of the study is to evaluate the effect of ORM-12741 on receptor occupancy by positron emission tomography with different doses and plasma concentrations. The pharmacokinetic profile and safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Good general health ascertained by detailed medical history and physical examination
* Males between 18 and 45 years
* Body mass index (BMI; weight/height2) between 18-30 kg/m2
* Weight 55-95 kg

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastro-intestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator
* Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant medication during the study
* Regular consumption of more than 21 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol).
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day
* Inability to refrain from using nicotine-containing products during the stay at the study centre
* Inability to refrain from consuming caffeine-containing beverages during the stay at the study centre e.g. propensity for headache when refraining from caffeine-containing beverages
* Blood donation or loss of significant amount of blood within 3 months prior to the screening visit
* Abnormal 12-lead electrocardiogram (ECG) finding of clinical relevance
* Any abnormal value of laboratory, vital signs, or physical examination, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk for the subject if he takes part into the study
* Anatomical abnormality in brain MRI which may in the opinion of the investigator interfere with the interpretation of the PET results
* Participation in another clinical drug study within 3 months prior to the start of this study or earlier participation in a clinical study with ORM-12741
* Participation in a prior PET study
* Any contraindication to MRI of the brain

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Receptor occupancy | 1 day

SECONDARY OUTCOMES:
Pharmacokinetic variables including peak concentration in plasma, time to peak concentration, area under the plasma concentration-time curve | 1 day
Safety variables including blood pressure, heart rate, electrocardiogram, physical examination, laboratory safety variables (haematology, chemistry, serology, urinanalysis) and adverse events. | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, MD, PhD, Principal Investigator — Turku PET Centre
Locations (1):
- Turku PET centre, Turku, Finland

REFERENCES:
- [Derived] Shahid M, Rinne JO, Scheinin M, Virta J, Marjamaki P, Solin O, Arponen E, Sallinen J, Kuokkanen K, Rouru J. Application of the PET ligand [11C]ORM-13070 to examine receptor occupancy by the alpha2C-adrenoceptor antagonist ORM-12741: translational validation of target engagement in rat and human brain. EJNMMI Res. 2020 Dec 9;10(1):152. doi: 10.1186/s13550-020-00741-y. PMID 33296042